CLINICAL TRIAL: NCT01893190
Title: Nimodipine Microparticles to Enhance Recovery While Reducing TOxicity After subarachNoid Hemorrhage: Phase I/IIa Multicenter, Controlled, Randomized, Open Label, Dose Escalation, Safety, Tolerability, and Pharmacokinectic Study Comparing EG-1962 and Nimodipine in Patients With Aneurysmal Subarachnoid Hemorrhage
Brief Title: Safety and Tolerability Study of EG-1962 in Aneurysmal Subarachnoid Hemorrhage
Acronym: NEWTON
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Edge Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EG-01-1962-02; 2013-000954-23 (EudraCT Number)
Record Dates: First submitted 2013-07-02; First posted 2013-07-08 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Ruptured Cerebral Aneurysm; Ruptured Berry Aneurysm
Keywords: Ruptured saccular aneurysm; nimodipine; safety; tolerability; Subarachnoid hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Nimodipine; EG-1962

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nimodipine (Active Comparator): Nimodipine 60mg q4h for 21 days - oral
  Interventions: Drug: Nimodipine
- Nimodipine Microparticles (Experimental): Single intraventricular injection
  Interventions: Drug: Nimodipine Microparticles

INTERVENTIONS:
Drug: Nimodipine — Based upon Investigator Judgement
  Other Names: Nimodipine Softgel; Nimodipine Tablet
  Arms: Nimodipine
Drug: Nimodipine Microparticles — Based upon Investigator Judgement
  Other Names: EG-1962
  Arms: Nimodipine Microparticles

SUMMARY:
Phase 1/2a Multicenter, Controlled, Randomized, Open Label, Dose Escalation, Safety, Tolerability, and Pharmacokinetic Study Comparing EG-1962 and Nimodipine in Patients with Aneurysmal Subarachnoid Hemorrhage

DETAILED DESCRIPTION:
This is a Phase 1/2a multicenter, controlled, open label, and randomized, study.

Part 1 of the study is a single dose escalation period to determine the MTD of EG-1962. During this period, a maximum of 6 dose level cohorts with up to 12 patients per cohort will be enrolled. In each cohort, patients will be randomly assigned in a ratio of 3:1 to receive either intraventricular EG 1962 or enteral nimodipine, respectively. The first cohort will receive 100 mg EG 1962. Upon completion of the dose escalation period, a safe and tolerable dose will be selected for further study.

Part 2 of the study is a treatment period to assess the safety and tolerability of the selected dose of EG-1962.

The safety and tolerability of a single intraventricular dose of EG 1962 will be compared to enteral nimodipine (60 mg given every 4 hours orally or via nasogastric or gastrostomy tube) for 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18 to 75 years, inclusive;
* WFNS Grade 2, 3, or 4 assessed after treatment of the aneurysm but prior to administration of EG-1962;
* Ruptured saccular aneurysm confirmed by angiography (catheter or CTA) and treated by neurosurgical clipping or endovascular coiling;
* Subarachnoid hemorrhage on baseline CT scan that is diffuse (clot present in both hemispheres) thick (>4 mm) or thin, or local thick;
* External ventricular drain (EVD) in place;
* The patient is able to receive EG-1962 within 60 hours of the onset of subarachnoid hemorrhage (SAH). Onset of SAH is defined as the time the patient experiences the first symptom of SAH (e.g., severe headache or loss of consciousness reported either by patient or by a witness). If found unconscious, the onset of SAH is defined as the last time the patient was seen at baseline neurological state;
* Weight >45 kg;
* Hemodynamically stable after resuscitation with systolic blood pressure (SBP) ≥90 mm Hg without the use of inotropic agents;
* Signed informed consent from the patient or the patient's legal representative after the completion of aneurysm repair and after all study criteria are confirmed; and
* Female patients of child bearing potential must have negative pregnancy test . Male patients must agree to use adequate birth control during the study and up to 1 month after the discontinuation of the study drug treatment.

Exclusion Criteria:

* Subarachnoid hemorrhage due to causes other than a saccular aneurysm (e.g., trauma or rupture of fusiform or infective aneurysm);
* WFNS Grade 1 or 5 assessed after completion of the aneurysm repair but prior to administration of EG-1962;
* Increased intracranial pressure >30 mm Hg in sedated patients lasting >4 hours anytime since admission;
* Intraventricular or intracerebral hemorrhage in absence of SAH or with only local, thin SAH;
* Angiographic vasospasm prior to aneurysm repair procedure, as documented by catheter angiogram or CT angiogram;
* Major complication during aneurysm repair such as, but not limited to, massive intraoperative hemorrhage, brain swelling, arterial occlusion, or inability to secure the ruptured aneurysm;
* Aneurysm repair requiring flow diverting stent or stent-assisted coiling and dual antiplatelet therapy;
* Hemodynamically unstable prior to administration of study drug (i.e., SBP <90 mm Hg, requiring >6 L colloid, or crystalloid fluid resuscitation;
* Cardiopulmonary resuscitation was required following SAH;
* Female patients with positive pregnancy test (blood or urine) at screening;
* History within the past 6 months and/or physical finding on admission of decompensated heart failure (New York Heart Association Class III and IV or heart failure requiring hospitalization);
* Acute myocardial infarction within 3 months prior to the administration of the study drug;
* Symptoms or electrocardiogram (ECG)-based signs of acute myocardial infarction or unstable angina pectoris on admission;
* Electrocardiogram evidence and/or physical findings compatible with second or third degree heart block or of cardiac arrhythmia associated with hemodynamic instability;
* Echocardiogram, if performed as part of standard-of-care before treatment, revealing a left ventricular ejection fraction <40%;
* Severe or unstable concomitant condition or disease (e.g., known significant neurologic deficit, cancer, hematologic, or coronary disease), or chronic condition (e.g., psychiatric disorder), that, in the opinion of the Investigator, may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results;
* Patients who have received an investigational product or participated in another interventional clinical study within 30 days prior to randomization. Patients participating in a non-interventional study that has no bearing on assessment of EG-1962 or enteral nimodipine can be enrolled per guidelines of the local Institutional Review Board (IRB) / independent Ethics Committee (IEC).
* Kidney disease as defined by plasma creatinine ≥2.5 mg/dl (221 μmol/l); liver disease as defined by total bilirubin >3 mg/dl (51.3 μmol/l); and/or known diagnosis or clinical suspicion of liver cirrhosis; or Known hypersensitivity to nimodipine or other dihydropyridine calcium channel antagonists, poly-D, L-lactide-co-glycolide (PLGA), or hyaluronic acid.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2013-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Dose Escalation Period | 3 Months
  To determine the maximum tolerated dose (MTD) of intraventricular EG 1962.

SECONDARY OUTCOMES:
PK measurements | 3 Months
  To measure plasma and cerebrospinal fluid (CSF) concentrations of nimodipine

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hanggi, Principal Investigator — HHU
Locations (23):
- United States (16):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Rush University Medical Center, Chicago, Illinois
  - University of Maryland Medical Cnter, Baltimore, Maryland
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Overlook Medical Center, Summit, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Mount Sinai Medical Center, New York, New York
  - Columbia University, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Mayfield Clinic Inc, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
- Canada (5):
  - University of Calgary, Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network - Toronto General Division, Toronto Western Hospital, Toronto, Ontario
  - University of Saskatchewan, Royal University Hospital, Saskatoon, Saskatchewan
- Charles University, Department of Neurosurgery, Prague, Czechia
- Helsinki University Central Hospital, Helsinki, Finland

REFERENCES:
- [Derived] Macdonald RL, Hanggi D, Strange P, Steiger HJ, Mocco J, Miller M, Mayer SA, Hoh BL, Faleck HJ, Etminan N, Diringer MN, Carlson AP, Aldrich F; NEWTON Investigators. Nimodipine pharmacokinetics after intraventricular injection of sustained-release nimodipine for subarachnoid hemorrhage. J Neurosurg. 2019 Dec 6;134(1):95-101. doi: 10.3171/2019.9.JNS191366. Print 2021 Jan 1. PMID 31812149
- [Derived] Hanggi D, Etminan N, Aldrich F, Steiger HJ, Mayer SA, Diringer MN, Hoh BL, Mocco J, Faleck HJ, Macdonald RL; NEWTON Investigators. Randomized, Open-Label, Phase 1/2a Study to Determine the Maximum Tolerated Dose of Intraventricular Sustained Release Nimodipine for Subarachnoid Hemorrhage (NEWTON [Nimodipine Microparticles to Enhance Recovery While Reducing Toxicity After Subarachnoid Hemorrhage]). Stroke. 2017 Jan;48(1):145-151. doi: 10.1161/STROKEAHA.116.014250. Epub 2016 Dec 8. PMID 27932607
- [Derived] Hanggi D, Etminan N, Macdonald RL, Steiger HJ, Mayer SA, Aldrich F, Diringer MN, Hoh BL, Mocco J, Strange P, Faleck HJ, Miller M. NEWTON: Nimodipine Microparticles to Enhance Recovery While Reducing Toxicity After Subarachnoid Hemorrhage. Neurocrit Care. 2015 Oct;23(2):274-84. doi: 10.1007/s12028-015-0112-2. PMID 25678453